CLINICAL TRIAL: NCT05898893
Title: Prospective, Multi-Center, Open-Label, Single-Arm Registration Trial Of The Tubridge Plus For The Treatment Of Wide-Necked Intracranial Aneurysms
Brief Title: PARAT PLUS (The Tubridge Plus For The Treatment Of Wide-Necked Intracranial Aneurysms)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MicroPort NeuroTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TB2-2021-01-0A
Record Dates: First submitted 2023-05-11; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Device: Microport NeuroTech Tubridge Plus flow-diverter Stent

INTERVENTIONS:
Device: Microport NeuroTech Tubridge Plus flow-diverter Stent — Intracranial stent for wide-necked aneurysms

SUMMARY:
A trial to evaluate the safety and efficacy of the Tubridge Plus flow-diverter stent for the treatment of intracranial wide-necked aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old (as of the date of signing the informed consent form);
2. CTA, MRA or DSA angiography diagnosed as a large intracranial carotid artery or vertebral artery aneurysm (largest diameter of the aneurysm >= 10mm) or medium to small aneurysms (maximum diameter <10mm) (including saccular aneurysms and recurrent saccular aneurysms);
3. The neck of aneurysm 4mm or the body-to-neck ratio of aneurysm < 2;
4. The diameter of the parent vessel is 2.0mm-6.5mm;
5. Subjects who are suitable for treatment with Tubridge Plus flow-diverted dense mesh stent alone or in combination with coils;
6. Subjects are willing to follow up and evaluate according to the requirements of the clinical trial protocol;
7. The subjects or their guardians can understand the purpose of the trial, participate voluntarily and sign the informed consent.

Exclusion Criteria:

1. Aneurysm related to AVM and MMD;
2. Ruptured aneurysm within 30 days;
3. Multiple aneurysms;
4. Subjects with significant stenosis (stenosis rate >= 50%) or occlusion of parent artery
5. Recurrent aneurysms after stent or stent-assisted coil embolization;
6. Subjects with morphologies or lesions that may interfere with device use, including but not limited to: carotid artery dissection, vasculitis, Aortic dissection, restriction of vascular access (such as severe intracranial vascular tortuosity, severe intracranial vasospasm and no response to drug therapy, obstruction of device access due to other anatomical or clinical lesions);
7. Subjects who are not suitable for anesthesia or endovascular treatment, such as severe diseases of the heart, lung, liver, spleen, and kidney, brain tumors, severe active infection, disseminated intravascular coagulation, and a history of severe mental illness;
8. Subjects who underwent or plan undergo to major surgical operations (such as implantation of internal fixation devices for extremity fractures, tumor resection, major organ surgery, etc.) within 30 days before signing the informed consent form or 60 days after signing the informed consent form;
9. Modified Rankin score >= 4 points ;
10. The life expectancy of the subjects is less than 12 months;
11. Subjects who have participated in clinical trials of other drugs or medical devices before enrollment and did not reach the end point.
12. The researchers judged that the subjects had poor compliance and could not complete the study as required;
13. Subjects with suspected history of allergy to nickel-titanium, platinum, platinum-iridium alloys and other materials;
14. Subjects who cannot receive antiplatelet aggregation or anticoagulation therapy;
15. Subjects have or may have had a serious reaction to the contrast agent and could not complete the pre-treatment medication;
16. Women who are pregnant or breastfeeding;
17. Other conditions deemed inappropriate by the investigator to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Complete occlusion（Raymond I） rate of aneurysm at 6 months after procedures | 6months±30 days
  Complete occlusion（Raymond I） rate of aneurysm at 6 months after procedures

SECONDARY OUTCOMES:
Complete occlusion（Raymond I） rate of aneurysm at 12 months after procedures | 12months±60 days
  Complete occlusion（Raymond I） rate of aneurysm at 12 months after procedures
Successful treatment（Raymond I or II）rate of aneurysm at 6 months after procedures | 6months±30 days
  uccessful treatment（Raymond I or II）rate of aneurysm at 6 months after procedures
Successful treatment（Raymond I or II）rate of aneurysm at 12 months after procedures | 12months±60 days
  Successful treatment（Raymond I or II）rate of aneurysm at 12 months after procedures
Retreatment rate of target aneurysm during follow-up | 12months±60 days
  Retreatment rate of target aneurysm during follow-up
Success rate of stent implantation | Immediate evaluation after intervention
  Success rate of stent implantation
The proportion of subjects with ipsilateral stroke or neurogenic death to their target aneurysm at 1 month postoperatively, 6 months postoperatively, and 1 year postoperatively; | 12months±60 days
  The proportion of subjects with ipsilateral stroke or neurogenic death to their target aneurysm at 1 month postoperatively, 6 months postoperatively, and 1 year postoperatively;
The proportion of subjects with in-stent stenosis (stenosis ≥50% and <100%) within 6 months after procedures | 6months±30 days
  The proportion of subjects with in-stent stenosis (stenosis ≥50% and <100%) within 6 months after procedures
Proportion of subjects with complete in-stent occlusion within 6 months after procedures | 6months±30 days
  Proportion of subjects with complete in-stent occlusion within 6 months after procedures
Device-related adverse events, serious adverse events within 1 month, 6 months, and 1 year after procedures | 12months±60 days
  Device-related adverse events, serious adverse events within 1 month, 6 months, and 1 year after procedures

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, Principal Investigator — Changhai Hospital
Locations (8):
- China (8):
  - West China Hospital of Sichuan University, Chendu
  - Huashan Hospital of Fudan University, Shanghai
  - Shanghai Changhai Hospital, Shanghai
  - Clinical Research Ethics Committee of Shenzhen Second People's Hospital, Shenzhen
  - Zhongnan Hospital, Wuhan University, Wuhan
  - The Second Affiliated Hospital of PLA Air Force Military Medical University, Xi'an
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Zhujiang Hospital,Southern Medical University, Zhujiang

IPD SHARING:
Plan to Share IPD: No